CLINICAL TRIAL: NCT00501202
Title: A Randomized, Double-Blind, Placebo-Controlled, Crossover Study of RWJ 333369 for the Treatment of Neuropathic Pain in Diabetic Peripheral Neuropathy.
Brief Title: Study for Safety and Effectiveness of RWJ-333369 (Carsibamate) for the Treatment of Diabetic Peripheral Neuropathy (DPN).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR010366; 333369NPP2002
Record Dates: First submitted 2007-07-12; First posted 2007-07-16 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Diabetic Neuropathy, Painful; Diabetic Neuralgia; Diabetic Polyneuropathy; Diabetic Mononeuropathy
Keywords: diabetes mellitus; diabetic microvascular injury; painful polyneuropathy.
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus | interventions — S-2-O-carbamoyl-1-o-chlorophenyl-ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 002 (Placebo Comparator): placebo twice daily for 4 weeks
  Interventions: Drug: placebo
- 001 (Experimental): RWJ-333369 (carisbamate) 200 mg tablet twice daily for 4 weeks
  Interventions: Drug: RWJ-333369 (carisbamate)

INTERVENTIONS:
Drug: placebo — twice daily for 4 weeks
  Arms: 002
Drug: RWJ-333369 (carisbamate) — 200 mg tablet twice daily for 4 weeks
  Arms: 001

SUMMARY:
The purpose of this study is to evaluate the safety, effectiveness, and tolerability of 200 mg of RWJ-333369 given twice daily by mouth compared with placebo in the treatment of Diabetic Peripheral Neuropathy (DPN).

DETAILED DESCRIPTION:
Diabetes mellitus is the most common cause of neuropathy in the Western World, with up to 50% of patients developing neuropathy as a long-term complication of the illness, of whom 10% experience pain. Diabetic neuropathy most often affects the lower extremities and may be severe if inadequately treated. Blood glucose control is a critical treatment element, and several medications have been demonstrated to be effective in treating Diabetic Peripheral Neuropathy (DPN), including antiepileptic drugs, antidepressants and opioid analgesics. These medications are often limited by incomplete pain relief and side effects. This is a randomized (study medication is assigned by chance), double-blind (neither the Investigator or the patient know the name of the assigned study medication), placebo-controlled, crossover, parallel-group, multicenter study to determine the effectiveness and safety of 200 mg of RWJ-333369 given twice daily by mouth for 4 weeks compared with placebo in patients with DPN. The study hypothesis is that 200 mg of RWJ-333369 given twice daily by mouth for 4 weeks will be more effective than placebo in reducing pain due to DPN, as measured by average daily DPN pain scores. Patients will receive 200 mg of RWJ-333369 or matching placebo tablets, given in equally divided doses twice daily by mouth with or without food, for 4 weeks in each of the 2 treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Have diabetes mellitus (Type 1 or 2) for longer than 1 year
* Have clinical evidence of diabetic peripheral neuropathy in the lower extremities for 1 to 5 years before study entry
* Experienced lower extremity pain due to diabetic peripheral neuropathy on nearly a daily basis for the previous 3 months
* Have hemoglobin A1c levels less than or equal to 10%
* Have a stable diabetic treatment regimen, including oral medications for controlling diabetes, insulin, or diet for 3 months before screening
* Women must be postmenopausal for at least 2 years, sexually abstinent, or if sexually active, be practicing an effective method of birth control, and have a negative serum pregnancy test at screening.

Exclusion Criteria:

* History of a poor response to 3 or more medications for diabetic peripheral neuropathy (DPN), with poor response is defined as treatment with medications in the following categories of therapy for at least 1 month at therapeutic dosages without at least moderate improvement, as judged by the study doctor: antiepileptic drugs, tricyclic antidepressants, serotonin norepinephrine reuptake inhibitors (SNRIs), opioid analgesics, or lidocaine patch
* currently taking tricyclic antidepressants, Coumadin (warfarin), or continued treatment with an antiepileptic drug for any indication, Note: If taking these medications, to be eligible for the study, they must be tapered and discontinued
* Prior neurolytic treatment (destruction of nerves by the application of chemicals, heat, or cold), intrathecal pumps, or spinal cord stimulators for DPN pain
* Use of herbal creams or ointments for pain relief within 48 hours, capsaicin within 6 months, or systemic corticosteroids within 3 months before the baseline period
* Prior exposure to RWJ-333369 (carisbamate).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2007-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The mean of the last 7 average daily DPN scores of the first treatment period on days when study drug is taken. | 4 weeks

SECONDARY OUTCOMES:
The means of the last 7 average daily DPN pain scores with no use of rescue medication, the last 7 current daily DPN pain scores, the last 7 maximum daily DPN pain scores, and the last 7 daily sleep interference scores. | 4 weeks (2 four-week treatment periods (crossover design)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.